CLINICAL TRIAL: NCT00736138
Title: Effect of Training and Pellots in Treatment of Foot Pain Caused by Hyperpronation
Brief Title: Hyperpronation and Foot Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northern Orthopaedic Division, Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ON-02-001-OSi
Record Dates: First submitted 2008-08-14; First posted 2008-08-15 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: Arthritis of Knee

ARMS (2):
- 1 (Active Comparator): training and pellots
  Interventions: Procedure: training and pellots
- 2 (No Intervention): control

INTERVENTIONS:
Procedure: training and pellots — training and pellots
  Arms: 1

SUMMARY:
Effects of training and pellots

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

-

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-06; Primary Completion 2013-04 (Actual); Study Completion 2013-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ole H Simonsen, MD, Principal Investigator — Northern Orthopaedic Division
Locations (1):
- Northern Orthopaedic Division, Klinik Aalborg, Aalborg, Northern Jutland, Denmark